CLINICAL TRIAL: NCT05065021
Title: Re-VOLVE: A Phase II Clinical Trial in Women With Ovarian Cancer Progressing Post-PARP Inhibitor With Treatment Adapted to Real-time Assessment of Evolving Genomic Resistance
Brief Title: Using Genetic Profile to Determine the Treatment for Patients With Ovarian Cancer Who Previously Received a PARP-inhibitor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Re-VOLVE; 21-5915 (Other: University Health Network)
Record Dates: First submitted 2021-09-29; First posted 2021-10-01 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer; High Grade Serous Cancer; High Grade Endometrioid Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — niraparib; dostarlimab; Bevacizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Initial/Cohort C (Experimental): Niraparib by mouth (orally), once a day, every day. Bevacizumab, by vein (intravenously), once every 3 weeks for up to 1 year, then every 6 weeks.
  Interventions: Drug: Niraparib; Drug: Bevacizumab
- Cohort A (Experimental): Niraparib by mouth (orally), once a day, every day. Bevacizumab, by vein (intravenously), once every 3 weeks for up to 1 year, then every 6 weeks.
  Dostarlimab, by vein (intravenously), once every 3 weeks for 4 doses, then every 6 weeks afterwards.
  Interventions: Drug: Niraparib; Drug: Dostarlimab; Drug: Bevacizumab
- Cohort B (Experimental): Paclitaxel, by vein (intravenously), once a week. Bevacizumab, by vein (intravenously), once every 3 weeks for up to 1 year, then every 6 weeks.
  Dostarlimab, by vein (intravenously), once every 3 weeks for 4 doses, then every 6 weeks afterwards.
  Interventions: Drug: Dostarlimab; Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Niraparib — Niraparib works by blocking poly(ADP-ribose) polymerases (PARP) 1 and PARP 2 from working. PARP 1 and PARP 2 are proteins that are involved in cell growth, cell survival, and cell death, including cancer cells. It is believed that blocking PARP1 and PARP 2 from working will slow or stop the growth of cancer cells.
  Other Names: ZEJULA
  Arms: Cohort A; Initial/Cohort C
Drug: Dostarlimab — Dostarlimab is a monoclonal antibody. Antibodies are proteins that are naturally found in the blood stream that fight infections. A monoclonal antibody is a special kind of antibody that is created in a laboratory that seeks out specific proteins in the body that may be involved in cancers to stop tumor growth. Dostarlimab attaches to PD-1 and inhibits the interaction of PD-L1 and PD-L2 with PD-1.
  Arms: Cohort A; Cohort B
Drug: Bevacizumab — Bevacizumab is a chemotherapy drug commonly used for the treatment of various cancers.
Drug: Paclitaxel — Paclitaxel is a chemotherapy drug commonly used for the treatment of various cancers.
  Arms: Cohort B

SUMMARY:
The purpose of this research study is to see how useful it is to look at biomarkers in the blood and tumor tissue of participants with ovarian, fallopian tube or primary peritoneal cancer who have previously received treatment with a drug called a PARP inhibitor, and using the results to determine the best treatment for these participants. Biomarkers are molecules such as genes (molecules that contain instructions for the development and function of cells in the body) and proteins that may be used to see how well a body responds to certain treatments.

DETAILED DESCRIPTION:
Participants who join the study will first have samples of their blood and tumor tissue collected for biomarker testing. The testing will involve a method called "sequencing". This test will look for changes in the genes of your tumor. The results of the testing will be what is called the participant's molecular profile.

All participants will first receive bevacizumab and niraparib for 3 cycles. A cycle will be 21-days in length.

Once the participant's molecular profile has been determined, the study doctor will discuss the results with the participants and they may be referred to a genetic counsellor.

Participants will then be assigned to a study cohort (group) and receive a combination of the study drugs based on the results of their genetic testing:

* Cohort A: Participants who do not have the required gene changes will be assigned to receive niraparib, bevacizumab, and dostarlimab
* Cohort B: Participants who have certain gene changes will receive paclitaxel, bevacizumab, and dostarlimab.
* Cohort C: If the participant and the study doctor think that the participant is benefitting from the combination of bevacizumab and niraparib, or the molecular profile shows that bevacizumab and niraparib is the most suitable, the participant may continue to receive this drug combination.

Participants will receive the study drug combination until disease worsening or they meet the criteria for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Histologically confirmed ovarian, fallopian tube or primary peritoneal cancer, high grade serous or high grade endometrioid histology subtype.
* Patients must have relapsed disease, either platinum-sensitive, resistant or refractory, with no limit to number of lines of prior systemic therapy.
* Radiographically documented disease progression within 28 days of registration.
* Patient must have measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
* Progression on any prior Poly (ADP-ribose) polymerase (PARP) inhibitor therapy, with no limit to number of prior lines of PARP inhibitors.
* Patients must have adequate bone marrow, renal and hepatic function within 7 days of registration
* Left ventricular ejection fraction (LVEF) > 50% by echocardiograms or multigated acquisition (MUGA) scan within 28 days of registration.
* Patients are willing to undergo tumor biopsy pre-treatment (tissue at the time of progression on PARP inhibitor therapy).
* Availability of archival tissue (prior to PARP inhibitor therapy) for analysis.
* Women of child-bearing potential must agree to use a highly effective contraceptive method for study-required period. A negative high sensitive urine or serum pregnancy test within 3 days prior to the initiation of therapy will be required for women of childbearing potential.
* Patient must agree to not donate blood during the study or for 90 days after the last dose of study treatment.
* Patient must agree to not breastfeed during the study or for 30 days after the last dose of study treatment.

Exclusion Criteria:

* Treatment with an investigational (other than PARP inhibitor) drug within 30 days and treatment with PARP inhibitor within 14 days prior to the first dose of study medication.
* Major surgery within 4 weeks of registration or ongoing clinically significant post-surgical complications.
* Patients with current or are at high-risk of developing fistula, or any other gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients with current or history of bowel obstruction within the last 3 months.
* Untreated unstable brain or leptomeningeal metastases.
* Greater than +1 proteinuria on two consecutive dipsticks within 14 days of registration.
* Unresolved toxicity of > grade 1 from previous anti-cancer therapy (including radiotherapy).

.History of poorly controlled hypertension or resting blood pressure >140/90 mmHg in the presence or absence of a stable regimen of anti-hypertensive therapy within 7 days of registration.

* Mean QTc >470 msec in screening electrocardiograms within 7 days of registration or history of familial long QT syndrome.
* Any evidence of severe or uncontrolled diseases such as but not limited to unstable or uncompensated respiratory, cardiac, hepatic, renal disease or psychiatric illness/social situations that would limit compliance with study requirements.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, paclitaxel, dostarlimab, or niraparib.
* Patients who have received prior weekly paclitaxel in the recurrent ovarian cancer setting.
* Patients who have received prior PD-1 inhibitor for ovarian cancer.
* Active autoimmune disease that has required systemic treatment in the past 2 years.
* History of interstitial lung disease.
* Patients with myelodysplastic syndrome/acute myeloid leukemia
* Previous allogenic bone marrow transplant.
* Immuno-compromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV), patients with known active hepatitis (i.e., hepatitis B or C).
* Patients with significant hemorrhage (>30 mL bleeding/episode in previous 3 months) or hemoptysis (>5 mL fresh blood in previous 4 weeks).
* Patients who have had recent (within 2 weeks of registration, or until any wound has completely healed) major thoracic or abdominal surgery prior to study start, or a surgical incision that is not fully healed.
* History of stroke or transient ischemic attack within six months.
* Patients that are receiving other anti-cancer therapy (except patient currently progressing on treatment with PARP inhibitor), radiotherapy, biological therapy or other novel agent prior to start of study treatment.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the participant inappropriate for entry into the study.
* History of other primary second malignancies (except for adequately treated cutaneous basal or squamous cell carcinoma or carcinoma in situ) within < 3 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-06-06 (Estimated); Study Completion 2025-06-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants that achieve biomarker-guided treatment | 3 years
Response rate percentage | 3 years

SECONDARY OUTCOMES:
Overall response rate for Cohort A | 3 years
Overall response rate for Cohort B | 3 years
Overall response rate for initial cohort/Cohort C | 3 years
Progression-free survival rate for initial cohort/Cohort C | 3 years
Progression-free survival rate for initial cohort/Cohort A | 3 years
Progression-free survival rate for initial cohort/Cohort B | 3 years
CA125 response rate for initial cohort/Cohort C | 3 years
CA125 response rate for Cohort A | 3 years
CA125 response rate for Cohort B | 3 years
Disease control rate for initial cohort/Cohort C | 3 years
Disease control rate for Cohort A | 3 years
Disease control rate for Cohort B | 3 years
Percentage of participants with adverse events in the initial cohort/Cohort C | 3 years
Percentage of participants with adverse events in Cohort A | 3 years
Percentage of participants with adverse events in Cohort B | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada